CLINICAL TRIAL: NCT04933968
Title: Phase 1/2, Double-Blind, Placebo-Controlled, Dose Escalation and Expansion Study of ALVR106 in Addition to Standard of Care for the Treatment of High-Risk Patients With Respiratory Viral Infections After Hematopoietic Cell and Solid Organ Transplant
Brief Title: Study of ALVR106 in Patients With Respiratory Viral Infections After Hematopoietic Cell and Solid Organ Transplant
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Strategic sponsor decision
Sponsor: AlloVir (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: P-106-001
Record Dates: First submitted 2021-06-07; First posted 2021-06-22 (Actual); Results first posted 2024-06-06 (Actual); Last update posted 2024-06-06 (Actual); Status verified 2024-06

CONDITIONS: Respiratory Tract Viral Infections; Human Metapneumovirus (hMPV) Infection; Parainfluenza (PIV) Infection; Respiratory Syncytial Viral (RSV) Infection; Influenza Infection
Keywords: Respiratory virus; Hematopoietic Cell Transplant; Upper Respiratory Tract Infection; Bone Marrow Transplant; Human Metapneumovirus Infection; Parainfluenza; Respiratory Syncytial Virus (RSV); Multi-virus specific T cells (VST); Solid Organ Transplant (SOT)
MeSH Terms: conditions — Infections; Paramyxoviridae Infections; Respiratory Tract Infections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Placebo, visually identical to ALVR106
  Interventions: Biological: Placebo
- ALVR106 (Active Comparator): ALVR106, visually identical to placebo
  Interventions: Biological: ALVR106

INTERVENTIONS:
Biological: ALVR106 — Infusion, visually identical to placebo
  Arms: ALVR106
Biological: Placebo — Infusion, visually identical to ALVR106
  Arms: Placebo

SUMMARY:
A study to evaluate ALVR106; an allogeneic, off-the-shelf multi-virus specific T cell therapy that targets four community acquired respiratory viruses: respiratory syncytial virus (RSV), influenza, human metapneumovirus (hMPV), and/or parainfluenza virus (PIV) following hematopoietic cell transplant (HCT) and solid organ transplant (SOT).

DETAILED DESCRIPTION:
The study hypothesis is that the administration of ALVR106, multi-virus specific T cells, plus standard of care, to post HCT or SOT patients suffering from infection with any of the four targeted viruses (RSV, influenza, hMPV, and/or PIV) will be safe and demonstrate shorter time to resolution of the respiratory viral infection (as measured by resolution of symptoms and viral load clearance in nasal swab) compared to patients treated with placebo.

This trial will consist of two parts: Part A is Dose Escalation and Part B is Cohort Expansion.

ELIGIBILITY:
Inclusion Criteria:

* Undergone hematopoietic cell transplantation (HCT) ≥21 days or solid organ transplantation (SOT) ≥28 days prior to study treatment administration
* Detection of at least 1 target virus of interest (ie, RSV, influenza, hMPV, and/or PIV)
* Diagnosis of Upper or mild Lower Respiratory Tract Infection

Exclusion Criteria:

* Ongoing therapy with high-dose systemic corticosteroids (ie, prednisone equivalent dose >0.5 mg/kg/day)
* Infection by novel coronavirus disease 2019 (COVID-19)
* For HCT patients, evidence of Grade >2 GVHD; and for SOT patients, any history or evidence of GVHD

Ages: 17 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2022-03-21 (Actual); Primary Completion 2024-01-31 (Actual); Study Completion 2024-01-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (21):
- United States (21):
  - Scottsdale Healthcare Hospitals DBA HonorHealth, Scottsdale, Arizona
  - City of Hope, Duarte, California
  - University of Florida - Division of Hematology & Oncology, Gainesville, Florida
  - University of Miami - Sylvester Cancer Center, Miami, Florida
  - Northside Hospital, Atlanta, Georgia
  - University of Iowa, Iowa City, Iowa
  - University of Kansas Cancer Center, Kansas City, Kansas
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Roswell Park Comprehensive Cancer Center, Buffalo, New York
  - University of North Carolina - Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Wake Forest, Winston-Salem, North Carolina
  - The Cleveland Clinic Foundation, Cleveland, Ohio
  - Medical University of South Carolina, Charleston, South Carolina
  - Vanderbilt University Cancer Center, Nashville, Tennessee
  - Baylor College of Medicine, Houston, Texas
  - MD Anderson Cancer Center, Houston, Texas
  - MD Anderson, Houston, Texas
  - Virginia Commonwealth University, Richmond, Virginia
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
  - Froedtert Hospital and the Medical College of Wisconsin, Milwaukee, Wisconsin

REFERENCES:
- [Background] Vasileiou S, Turney AM, Kuvalekar M, Mukhi SS, Watanabe A, Lulla P, Ramos CA, Naik S, Vera JF, Tzannou I, Leen AM. Rapid generation of multivirus-specific T lymphocytes for the prevention and treatment of respiratory viral infections. Haematologica. 2020 Jan;105(1):235-243. doi: 10.3324/haematol.2018.206896. Epub 2019 Apr 19. No abstract available. PMID 31004020
- [Derived] Papayanni PG, Koukoulias K, Kuvalekar M, Watanabe A, Velazquez Y, Ramos CA, Leen AM, Vasileiou S. T cell immune profiling of respiratory syncytial virus for the development of a targeted immunotherapy. Br J Haematol. 2023 Aug;202(4):874-878. doi: 10.1111/bjh.18933. Epub 2023 Jun 15. PMID 37323051

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at study centers in the United States and participated from March 2022 until January 2024.
Pre-assignment Details: Participants with respiratory tract infections and clinical manifestations caused by respiratory syncytial virus, influenza virus, human metapneumovirus, and/or parainfluenza virus following hematopoietic cell or solid organ transplants were enrolled. Participants were randomized in a double-blind manner to receive placebo or one of four dose levels of ALVR106, from Dose A (lower dose) to Dose D (higher dose). Due to early study termination, no participants were enrolled into Part B.
Groups:
- Part A: Placebo: Participants were randomized to receive placebo, and were administered placebo as an intravenous (IV) infusion on Day 1. Participants returned to the clinic for assessments up to Day 14, and based on assessments could receive a second infusion of placebo on Day 14. Participants were followed for up to 12 months.
- Part A ALVR106 Cohort 1: Dose A: Participants were randomized to receive ALVR106, and were administered ALVR106 Dose A as an IV infusion on Day 1. Participants returned to the clinical site for assessments up to Day 14, and based on assessments could receive a second infusion of ALVR106 Dose A on Day 14. Participants were followed for up to 12 months.
- Part A ALVR106 Cohort 2: Dose B: Participants were randomized to receive ALVR106, and were administered ALVR106 Dose B as an IV infusion on Day 1. Participants returned to the clinical site for assessments up to Day 14, and based on assessments could receive a second infusion of ALVR106 Dose B on Day 14. Participants were followed for up to 12 months.
- Part A ALVR106 Cohort 3: Dose C: Participants were randomized to receive ALVR106, and were administered ALVR106 Dose C as an IV infusion on Day 1. Participants returned to the clinical site for assessments up to Day 14, and based on assessments could receive a second infusion of ALVR106 Dose C on Day 14. Participants were followed for up to 12 months.
- Part A ALVR106 Cohort 4: Dose D: Participants were randomized to receive ALVR106, and were administered ALVR106 Dose D as an IV infusion on Day 1. Participants returned to the clinical site for assessments up to Day 14, and based on assessments could receive a second infusion of ALVR106 Dose D on Day 14. Participants were followed for up to 12 months.
- Part B Expansion Cohort: It was planned to enroll and randomize participants at high-risk with upper respiratory tract infections into Part B to receive placebo or ALVR106 at the recommended Phase 2 dose (RP2D). Due to the early termination of the study, no participants were enrolled into the Part B expansion cohort.
Period: Overall Study
Arm/Group | Part A: Placebo | Part A ALVR106 Cohort 1: Dose A | Part A ALVR106 Cohort 2: Dose B | Part A ALVR106 Cohort 3: Dose C | Part A ALVR106 Cohort 4: Dose D | Part B Expansion Cohort
Started | 3 | 3 | 4 | 4 | 3 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 3 | 3 | 4 | 4 | 3 | 0
Not completed — Adverse Event | 0 | 0 | 1 | 1 | 0 | 0
Not completed — Lost to Follow-up | 1 | 0 | 1 | 0 | 0 | 0
Not completed — Randomized not treated | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Sponsor terminated study | 0 | 0 | 0 | 1 | 2 | 0
Not completed — Other | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Missing | 1 | 3 | 2 | 1 | 1 | 0

BASELINE CHARACTERISTICS:
Population: The modified intent-to-treat population for Part A which included all randomized participants who received any amount of ALVR106 or placebo and had confirmed virologic infection of interest at baseline (detectable viral load). One participant randomized to the placebo cohort did not receive study treatment and is not included. Due to early study termination, no participants were enrolled into Part B and therefore Part B is not included in the baseline analysis population.
Groups:
- Part A: Placebo: Participants were randomized to receive placebo, and were administered placebo as an IV infusion on Day 1. Participants returned to the clinic for assessments up to Day 14, and based on assessments could receive a second infusion of placebo on Day 14. Participants were followed for up to 12 months.
- Total: Total of all reporting groups
Arm/Group | Part A: Placebo | Part A ALVR106 Cohort 1: Dose A | Part A ALVR106 Cohort 2: Dose B | Part A ALVR106 Cohort 3: Dose C | Part A ALVR106 Cohort 4: Dose D | Total
Number analyzed (Participants) | 2 | 3 | 4 | 4 | 3 | 16
Age, Customized [Count of Participants; unit: Participants]
  ≤ 18 years | 0 | 0 | 0 | 0 | 0 | 0
  19 - 70 years | 2 | 3 | 4 | 4 | 3 | 16
  ≥ 71 years | 0 | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 2 | 3 | 1 | 1 | 7
  Male | 2 | 1 | 1 | 3 | 2 | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 1 | 1
  Not Hispanic or Latino | 2 | 3 | 4 | 4 | 2 | 15
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 1 | 3 | 4 | 4 | 3 | 15
  Not reported | 1 | 0 | 0 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs) (Part A)
Description: A TEAE was defined as an adverse event (AE) with a start date and time on or after the first dose of study treatment. A serious AE (SAE) was an AE that met at least one of the following serious criteria: fatal, life-threatening, requires in-patient hospitalization or prolongation of existing hospitalization; resulted in persistent or significant disability/incapacity; was a congenital anomaly/birth defect; or other important medical event. TEAEs of special interest (AESI) included new/worsening graft versus host disease, graft failure or rejection, cytokine release syndrome, infusion related reactions, new/worsening pneumonitis, and progressive dyspnea. Treatment-related refers to the assessment of a relationship between study treatment and the event by the investigator.
Time Frame: Day 1 up to 12 months
Population: The safety population included all randomized participants who received any amount of ALVR106 or placebo.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: Placebo | Part A ALVR106 Cohort 1: Dose A | Part A ALVR106 Cohort 2: Dose B | Part A ALVR106 Cohort 3: Dose C | Part A ALVR106 Cohort 4: Dose D
Number analyzed (Participants) | 2 | 3 | 4 | 4 | 3
Participants
  Any TEAE | 2 | 3 | 4 | 4 | 3
  Any treatment-related TEAE | 2 | 1 | 0 | 0 | 0
  Any AESI | 1 | 1 | 0 | 1 | 1
  Any treatment-related AESI | 1 | 0 | 0 | 0 | 0
  Any SAE | 0 | 2 | 3 | 3 | 1
  Any treatment-related SAE | 0 | 0 | 0 | 0 | 0
  Any TEAE leading to study treatment discontinuation | 0 | 0 | 0 | 0 | 0
  Any TEAE leading to death | 0 | 0 | 1 | 1 | 0

2. Primary Outcome: Change in Viral Load From Baseline to Day 28 (Part B)
Description: Change from Baseline in viral load as measured by quantitative PCR of nasal swab
Time Frame: Baseline and Day 28 (Part B)
Population: No participants were enrolled into Part B due to the early termination of the study.
Groups:
- Part B Expansion Cohort: It was planned to enroll and randomize participants at high-risk with upper respiratory tract infections into Part B to receive placebo or ALVR106 at the RP2D. Due to the early termination of the study, no participants were enrolled into the Part B expansion cohort.
Arm/Group | Part B Expansion Cohort
Number analyzed (Participants) | 0

3. Secondary Outcome: Identify the Recommended Phase 2 Dose (RP2D) (Part A)
Description: The RP2D was to be determined after the maximum tolerated dose was reached in Part A.
Time Frame: Day 1 up to 12 months
Population: All randomized participants who received ALVR106 in Part A.
Measure: Number; unit: x 10^5 cells/kg
Groups:
- All Doses ALVR106 (Part A): Participants who were randomized to receive ALVR106 in Part A, including Doses A, B, C, and D.
Arm/Group | All Doses ALVR106 (Part A)
Number analyzed (Participants) | 14
x 10^5 cells/kg | NA — The MTD and RP2D could not be determined due to too few dose-limiting toxicities during the study prior to early study termination.

4. Secondary Outcome: Change in Viral Load Cycle Threshold From Baseline to Day 28 (Part A)
Description: Viral load was measured by quantitative polymerase chain reaction (PCR) of nasal swab specimens. The cycle threshold value categorizes the concentration of viral genetic material in a participant's swab specimen, and the cycle threshold value represents the number of PCR cycles required to amplify the viral genetic material (as measured by fluorescence) to a detectable level that is distinguishable from baseline fluorescence, providing an estimate of viral load. Lower cycle threshold values indicate higher viral load and high values indicate lower viral load. A positive change from baseline indicates a decrease in the viral load. The baseline measurement was from a pre-dose nasal swab.
Time Frame: Baseline and Day 28
Population: The modified intent-to-treat population included all randomized participants who received any amount of ALVR106 or placebo and had confirmed virologic infection of interest at baseline (detectable viral load). Participants with baseline and Day 28 available data are included.
Measure: Mean (Standard Deviation); unit: cycles
Arm/Group | Part A: Placebo | Part A ALVR106 Cohort 1: Dose A | Part A ALVR106 Cohort 2: Dose B | Part A ALVR106 Cohort 3: Dose C | Part A ALVR106 Cohort 4: Dose D
Number analyzed (Participants) | 1 | 1 | 4 | 4 | 3
cycles | 8.60 (NA) — Standard deviation could not be determined as 1 participant was analyzed. | 4.40 (NA) — Standard deviation could not be determined as 1 participant was analyzed. | 8.43 (6.118) | 5.78 (4.696) | 7.47 (7.551)

5. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs) (Part B)
Time Frame: Day 1 up to 12 months
Population: No participants were enrolled into Part B due to the early termination of the study.
Arm/Group | Part B Expansion Cohort
Number analyzed (Participants) | 0

6. Secondary Outcome: Percentage Reduction in Viral Load From Baseline to Month 6 (Part B)
Time Frame: Day 1 and Month 6
Population: No participants were enrolled into Part B due to the early termination of the study.
Arm/Group | Part B Expansion Cohort
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Day 1 up to 12 months.
Description: AEs are presented for the safety population for Part A which included all randomized participants who received any amount of ALVR106 or placebo. Due to early study termination, no participants were enrolled into Part B and therefore Part B is not included in the AE data.
Arm/Group | Part A: Placebo | Part A ALVR106 Cohort 1: Dose A | Part A ALVR106 Cohort 2: Dose B | Part A ALVR106 Cohort 3: Dose C | Part A ALVR106 Cohort 4: Dose D
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/3 | 2/4 | 2/4 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/2 | 2/3 | 3/4 | 3/4 | 1/3
Other Adverse Events (participants affected / at risk) | 2/2 | 3/3 | 4/4 | 4/4 | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part A: Placebo (N=2) | Part A ALVR106 Cohort 1: Dose A (N=3) | Part A ALVR106 Cohort 2: Dose B (N=4) | Part A ALVR106 Cohort 3: Dose C (N=4) | Part A ALVR106 Cohort 4: Dose D (N=3)
Pneumonia (Infections and infestations) | NA | 1 | 0 | 0 | 0
COVID-19 (Infections and infestations) | NA | 1 | 0 | 0 | 0
Oesophageal candidiasis (Infections and infestations) | NA | 1 | 0 | 0 | 0
Odynophagia (Gastrointestinal disorders) | NA | 1 | 0 | 0 | 0
Acute myeloid leukaemia recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | NA | 0 | 2 | 0 | 0
Non-cardiac chest pain (General disorders) | NA | 0 | 1 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | NA | 0 | 1 | 0 | 0
Bronchial hyperreactivity (Respiratory, thoracic and mediastinal disorders) | NA | 0 | 1 | 0 | 0
Sepsis (Infections and infestations) | NA | 0 | 1 | 1 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | NA | 0 | 0 | 1 | 0
Liver function test increased (Investigations) | NA | 0 | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | NA | 0 | 0 | 1 | 1
Viral haemorrhagic cystitis (Infections and infestations) | NA | 0 | 0 | 1 | 0
Septic shock (Infections and infestations) | NA | 0 | 0 | 1 | 0
Small intestinal obstruction (Gastrointestinal disorders) | NA | 0 | 0 | 1 | 0
Pyrexia (General disorders) | NA | 0 | 0 | 1 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | NA | 0 | 0 | 0 | 1
Ascites (Gastrointestinal disorders) | NA | 0 | 0 | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | NA | 0 | 0 | 0 | 1
Hypervolaemia (Metabolism and nutrition disorders) | NA | 0 | 0 | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | NA | 0 | 0 | 0 | 1
Mental status changes (Psychiatric disorders) | NA | 0 | 0 | 0 | 1
Thyroiditis (Endocrine disorders) | NA | 0 | 0 | 0 | 1
Cardiomyopathy (Cardiac disorders) | NA | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part A: Placebo (N=2) | Part A ALVR106 Cohort 1: Dose A (N=3) | Part A ALVR106 Cohort 2: Dose B (N=4) | Part A ALVR106 Cohort 3: Dose C (N=4) | Part A ALVR106 Cohort 4: Dose D (N=3)
COVID-19 (Infections and infestations) | 1 | 0 | 3 | 0 | 0
Sepsis (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Oral candidiasis (Infections and infestations) | 0 | 0 | 0 | 0 | 2
Respiratory syncytial virus infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 1 | 1
BK virus infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0
COVID-19 pneumonia (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Clostridium difficile colitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Enterococcal bacteraemia (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Influenza (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Klebsiella bacteraemia (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Oesophageal candidiasis (Infections and infestations) | 0 | 0 | 0 | 0 | 0
Oral herpes (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Otitis media (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Parainfluenzae virus infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Rhinovirus infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Urinary tract infection enterococcal (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Vulvovaginal candidiasis (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1
Ascites (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Hyperaesthesia teeth (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Odynophagia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 1 | 0 | 1 | 1 | 1
Fatigue (General disorders) | 0 | 0 | 1 | 0 | 1
Non-cardiac chest pain (General disorders) | 1 | 0 | 0 | 0 | 0
Chills (General disorders) | 0 | 0 | 1 | 0 | 0
Influenza like illness (General disorders) | 0 | 0 | 0 | 1 | 0
Oedema peripheral (General disorders) | 0 | 0 | 1 | 0 | 0
White blood cell count decreased (Investigations) | 0 | 0 | 2 | 0 | 1
Neutrophil count decreased (Investigations) | 0 | 0 | 2 | 0 | 0
Platelet count decreased (Investigations) | 0 | 0 | 0 | 1 | 1
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 1 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 1 | 0
Blood bilirubin increased (Investigations) | 0 | 0 | 0 | 1 | 0
Blood creatine phosphokinase increased (Investigations) | 0 | 0 | 0 | 1 | 0
Blood creatinine increased (Investigations) | 0 | 0 | 1 | 0 | 0
Blood lactate dehydrogenase increased (Investigations) | 1 | 0 | 0 | 0 | 0
Transfer factor reduced (Investigations) | 0 | 0 | 1 | 0 | 0
Vitamin D decreased (Investigations) | 0 | 0 | 1 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0
Hypervolaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1
Vitamin B12 deficiency (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 2 | 0
Osteopenia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Myositis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1 | 0
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Hypercapnia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Sinus pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1 | 0
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0
Eosinophilia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0
Pancytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1
Ear pain (Ear and labyrinth disorders) | 0 | 1 | 1 | 0 | 0
Ear discomfort (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 1
Acute graft versus host disease in skin (Immune system disorders) | 1 | 0 | 0 | 1 | 0
Chronic graft versus host disease in lung (Immune system disorders) | 0 | 1 | 0 | 0 | 0
Chronic graft versus host disease oral (Immune system disorders) | 1 | 0 | 0 | 0 | 0
Post transplant lymphoproliferative disorder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0
Dizziness (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Encephalopathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Muscle tension dysphonia (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Paraesthesia (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 1 | 0
Hot flush (Vascular disorders) | 0 | 0 | 1 | 0 | 0
Superficial vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 1
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Hypogonadism (Endocrine disorders) | 0 | 0 | 0 | 0 | 1
Depression (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0
Polyuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1
Chimerism (Congenital, familial and genetic disorders) | 0 | 0 | 1 | 0 | 0
Dry eye (Eye disorders) | 0 | 0 | 1 | 0 | 0
Biliary obstruction (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1
Portal hypertension (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1

LIMITATIONS AND CAVEATS:
Results are included for Part A only as no participants were enrolled into Part B due to early study termination.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2022-05-19): https://cdn.clinicaltrials.gov/large-docs/68/NCT04933968/Prot_000.pdf
  • Statistical Analysis Plan (2022-02-25): https://cdn.clinicaltrials.gov/large-docs/68/NCT04933968/SAP_001.pdf